CLINICAL TRIAL: NCT00898209
Title: Serum and Exhaled Breath Condensate MALDI-MS of Lung Cancer
Brief Title: Serum and Exhaled Breath Condensate MALDI-MS of Lung Cancer. (SPORE)
Status: Terminated | Type: Observational
Why Stopped: This study competed with another VICC study
Sponsor: Vanderbilt-Ingram Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Pierre P. Massion, MD, Associate Professor of Medicine (Allergy, Pulmonary & Critical Care) and Cancer Biology; Pulmonary and Critical Care Medicine Doctor, Vanderbilt-Ingram Cancer Center
Other Study IDs: VICC THO 0332; VU-VICC-THO-0332; VU-VICC-030009
Record Dates: First submitted 2009-05-09; First posted 2009-05-12 (Estimated); Last update posted 2014-06-24 (Estimated); Status verified 2013-04

CONDITIONS: Lung Cancer
Keywords: stage I non-small cell lung cancer; stage II non-small cell lung cancer; stage IIIA non-small cell lung cancer; stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Peripheral blood lymphocyte DNA, and Exhaled breath condensate
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Health Volunteers: Blood and exhaled breath condensate will be collected.
  Interventions: Genetic: protein expression analysis; Genetic: proteomic profiling; Other: biologic sample preservation procedure; Other: laboratory biomarker analysis; Other: matrix-asst laser desorption/ionization time flight mass spectrometry; Other: questionnaire administration
- Patients at risk or already identified as having lung cancer: Blood and exhaled breath condensate will be collected.
  Interventions: Genetic: protein expression analysis; Genetic: proteomic profiling; Other: biologic sample preservation procedure; Other: laboratory biomarker analysis; Other: matrix-asst laser desorption/ionization time flight mass spectrometry; Other: questionnaire administration

INTERVENTIONS:
Genetic: protein expression analysis — Blood and exhaled breath condensate will be collected.
Genetic: proteomic profiling — Blood and exhaled breath condensate will be collected.
Other: biologic sample preservation procedure — Blood and exhaled breath condensate will be collected.
Other: laboratory biomarker analysis — Blood and exhaled breath condensate will be collected.
Other: matrix-asst laser desorption/ionization time flight mass spectrometry — Blood and exhaled breath condensate will be collected.
Other: questionnaire administration — Questionnaire will be completed.

SUMMARY:
RATIONALE: Collecting and storing samples of blood and exhaled breath from patients with cancer and from healthy participants to study in the laboratory may help doctors learn more about changes that occur in DNA and identify biomarkers related to cancer.

PURPOSE: This research study is collecting and analyzing samples of blood and exhaled breath from patients who have or are at high risk for lung cancer and from healthy participants.

DETAILED DESCRIPTION:
OBJECTIVES:

* To evaluate the ability of proteomic patterns in serum and exhaled breath condensate samples to detect and discriminate lung cancer from healthy and from high-risk individuals.
* To correlate proteomic patterns with tumor behavior.

OUTLINE: This is a multicenter study.

Blood and exhaled breath condensate samples are collected, whenever possible, at a time medically indicated for other purposes (e.g., work-up, pre-op, surgical procedures). The samples are used to produce genetic material (i.e., DNA, RNA) and molecular material (i.e., proteins) that will be stored for future studies, including studies that may not be related to lung cancer. Future genetic studies related to lung cancer may include studies of protein expression patterns via matrix-assisted laser desorption/ionization time of flight mass spectrometry that may serve as predictive molecular markers of lung cancer.

Participants complete a 15-minute Lung Spore Database questionnaire at the time of study enrollment to provide information on demographics (e.g., date of birth, address, phone number), medical and smoking history, personal and family history of cancer and cancer treatment, and current medications. Medical records are reviewed at the time of study enrollment and then over approximately 5 years to obtain information, including test results, associated with the diagnosis of cancer. Participants may also be contacted by phone at a later time to answer questions about their health status.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Meets 1 of the following criteria:

  * Normal healthy volunteer
  * At high risk for lung cancer (e.g., > 30-pack year history of smoking; chronic obstructive pulmonary disease; or disease-free after surgical resection of lung cancer)
  * Diagnosis of stage I, II, IIIA, IIIB, or IV lung cancer
* Must be willing to allow blood and exhaled breath condensate samples to be stored for genetic testing

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* Not specified

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy volunteers as well as patients at risk or already identified as having lung cancer.
Sampling Method: Non-Probability Sample
Enrollment: 564 (Actual)
Dates: Start 2003-04; Primary Completion 2009-02 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Ability of proteomic patterns to detect and discriminate lung cancer | Once at study entry
  Serum and exhaled breath condensate samples are collected from healthy and high-risk individual with lung cancer
Correlation of proteomic patterns with tumor behavior | Once at study entry

CONTACTS AND LOCATIONS:
Overall Officials: Pierre P. Massion, MD, Study Chair — Vanderbilt-Ingram Cancer Center